CLINICAL TRIAL: NCT05139706
Title: Montreal Database and Biorepository of Cancer Patients Treated With Immune Checkpoint Inhibitors for the Study of Immune-related Adverse Events
Brief Title: Montreal Immune-Related Adverse Events (MIRAE) Study
Acronym: MIRAE
Status: Recruiting | Type: Observational
Sponsor: Sir Mortimer B. Davis - Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Marie Hudson, MD, Marie Hudson, MD MPH FRCPC Principal Investigator, Rheumatologist, Division of Rheumatology and Department of Medicine, Jewish General Hospital and McGill University, Sir Mortimer B. Davis - Jewish General Hospital
Other Study IDs: MP-05-2019-1517
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Immune System Disorder; Inflammatory Reaction; Autoimmune Diseases
Keywords: irAEs; ICI (ICB); CTLA-4; PD-1; PDL-1; Pembrolizumab; Nivolumab; Ipilimumab; Cemiplimab; Atezolizumab; Avelumab; Durvalumab
MeSH Terms: conditions — Neoplasms; Immune System Diseases; Inflammation; Autoimmune Diseases; Diabetes Mellitus, Insulin-Dependent, 12

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Biospecimen Retention: Samples With DNA — * Whole blood
  * Peripheral blood mononuclear cells
  * Stool
  * Tissue biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Immune checkpoint inhibitors (ICI) are among the most promising approaches to fighting cancer. However, a substantial percentage of patients experience off-target adverse effects in the form of mild to severe inflammation in different organs, commonly called immune-related adverse events (irAEs). irAEs can lead to treatment discontinuation, or can be life-threatening in extreme cases. The causes of irAEs are largely unknown and there are no reliable predictive biomarkers. The Montreal Immune-Related Adverse Events (MIRAE) study collects clinical information and biospecimens (blood, tissue, stool) from cancer patients treated with ICI to facilitate research on the identification of predictive biomarkers of irAEs, their causes, and the design of effective management strategies.

DETAILED DESCRIPTION:
Background:

During cancer development and progression, cancer cells evolve to evade natural anti-tumor immunity. One major pathway of immune evasion involves the engagement of co-inhibitory receptors present on the surface of T cells that modulate their activation status, and therefore their ability to directly or indirectly kill tumor cells. These receptors are known as immune checkpoint inhibitors (ICI). Blockade of ICI using antibodies leads to prolonged T cell activation and unleashes the anti-tumor activity of T cells. ICI treatment for cancer has led to unprecedented advances in cancer treatment by prolonging survival of patients with previously refractory cancers. Among these ICI, CTLA-4, PD-1 and PDL-1 inhibitors have been shown to be effective cancer immunotherapies, and many other ICIs are now in pre-clinical and clinical development.

Although ICI cancer therapy is overall well tolerated, off-target immune reactions targeting healthy cells or tissues called immune-related adverse events (irAEs) develop in a substantial percentage of patients limiting the use of ICI therapy. irAEs target range from mild to severe and fatal. Currently, there are no reliable predictive biomarkers for the wide spectrum of irAEs and their clinical management in severe cases involves discontinuation of ICI therapy.

The Montreal Immune-Related Adverse Events (MIRAE) study is a biobank that collects human biological specimens (e.g., tissue, blood, plasma, PBMCs, saliva, stool) and the associated clinical information from cancer patients treated with ICI with the purpose of promoting research to identify clinical and biological predictors and mechanisms of irAEs, evaluate the effects of immunomodulatory treatment of irAEs on tumor biology, and investigate treatment strategies to minimize irAEs.

Objectives:

1. Identify biomarkers predictive of irAEs, including cellular, immunologic, genetic and microbial biomarkers; and
2. Evaluate the effects of immunomodulatory treatment of irAEs, and investigate treatment strategies that minimize irAEs and maximize ICI efficacy.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* cancer patients treated with ICI therapy (e.g., anti-CTLA-4, anti-PD-1, anti-PD-L1, and combinations)
* patients with primary autoimmune or autoinflammatory diseases that resemble immune-related adverse events (irAEs)
* healthy volunteers with non-inflammatory disorders, and without any history of cancer

Exclusion Criteria:

* Participants not able to provide informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer patients treated with ICI, patients with primary autoimmune or autoinflammatory diseases and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-01-21 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of immune-related adverse events | Up to 5 years
Biomarkers of irAE | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marie Hudson, MD, Principal Investigator — Jewish General Hospital, McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes